CLINICAL TRIAL: NCT03395951
Title: Clinical Observation of Mean Systemic Filling Pressure in Critical Care Patients With Continuous Diuretics Administration
Brief Title: Mean Systemic Filling Pressure Continuous Diuretics Critical Care Patients
Status: Completed | Type: Observational
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, L.P.B. Meijs, Principal investigator L.P.B. Meijs, MD, PhD-candidate Intensive Care Unit / resident cardiology, Catharina Ziekenhuis Eindhoven
Other Study IDs: n-WMO 2014-43
Record Dates: First submitted 2018-01-01; First posted 2018-01-10 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Sepsis; Heart Failure; Heart Diseases; Septic Shock; Surgery; Critically Ill
Keywords: Mean Systemic Filling Pressure; Diuretics; Pressure for venous return; Fluid Balance; De-escalation fluid therapy; De-resuscitation; Guyton; Guytonian Approach; Furosemide; Cardiac Output; Cardiac Index
MeSH Terms: conditions — Sepsis; Heart Failure; Heart Diseases; Shock, Septic; Critical Illness | interventions — Diuretics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Diuretics — Observation of hemodynamics during diuretics treatment within clinical indication.
  Other Names: Diuretic therapy

SUMMARY:
Within clinical settings observation of hemodynamic changes (e.g. mean systemic filling pressure, cardiac output) in critically ill patients with a clinical indication for deresuscitation with intravenous diuretic therapy.

DETAILED DESCRIPTION:
Rationale: The assessment of the cardiovascular state in critically ill patients is subject to difficulties in terms of the fact that several hemodynamic parameters, for example mean arterial blood pressure (MAP) and cardiac output (CO) supply insufficient information about the circulating volume and cardiac performance. There is a clinical need for adequate determination of intravascular volume status. However, in determining the intravascular fluid status of a patient, the lack of appreciation of the venous side of the circulation persists today, which is greatly due to the inability to appropriately assess the venous side of the circulation. The importance of the venous part of the circulation is moreover reflected by the fact that an increase in venous resistance does reduce CO many times more than a similar increase in arterial resistance. Mean systemic filling pressure (Pms), which is defined as the pressure equal to the pressure which would be measured if the heart should suddenly stop pumping and all (arterial and venous) the pressures in the entire circulatory system should be brought to equilibrium instantaneously, is a good, complete and reliable reflection of the total intravascular fluid compartment.

Positive fluid balance and /or substantial weight gain in critically ill patients is a common problem in the intensive care unit (ICU), potentially associated with a poor outcome. This problem, in association with hemodynamic instability and increase of creatinin, ureum and sodium, may lead to peripheral edema. Furosemide, a loop diuretic, is frequently administered to critically ill patients to increase urine output and to relieve edema.

Objective: Observing changes in Pms during continuous furosemide administration.

Study design: Prospective, observational study Study population: Patients with a PICCO® system with a positive fluid balance and / or substantial weight gain and therefore with a clinical indication for diuretic therapy.

Intervention: Continuous furosemide administration. Main study parameters/endpoints: Pms measured at baseline, changes in Pms during continuous furosemide administration.

Adverse events: No risks involved.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years
* PiCCO in situ (cardiac output device applied in light of clinical treatment)
* CVL in situ
* Clinical indication for continuous furosemide administration

Exclusion Criteria:

* Patients younger then 18 years
* Patients without PiCCO
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with a clinical indication for treatment with intravenous diuretics
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2014-10-01 (Actual); Study Completion 2015-01-31 (Actual)

PRIMARY OUTCOMES:
Change in mean systemic filling pressure (mmHg) | Baseline, every 5 minutes up to 30 minutes, 1 hour, 2 hours
  Decrease or increase in mean systemic filling pressure measured by bedside continuous hemodynamic monitor supplied with continuous cardiac output monitoring with PiCCO(R) device

SECONDARY OUTCOMES:
Change in cardiac index (L/min/m2) | Baseline, every 5 minutes up to 30 minutes, 1 hour, 2 hours
  Decrease/increase in cardiac index measured by bedside continuous hemodynamic monitor supplied with continuous cardiac output monitoring with PiCCO(R) device
Change in mean arterial pressure (mmHg) | Baseline, every 5 minutes up to 30 minutes, 1 hour, 2 hours
  Decrease/increase in mean arterial pressure measured by bedside continuous hemodynamic monitor supplied with continuous cardiac output monitoring with PiCCO(R) device
Change in central venous pressure (mmHg) | Baseline, every 5 minutes up to 30 minutes, 1 hour, 2 hours
  Decrease/increase in central venous pressure measured by bedside continuous hemodynamic monitor supplied with continuous cardiac output monitoring with PiCCO(R) device
Change in pressure for venous return (mmHg) | Baseline, every 5 minutes up to 30 minutes, 1 hour, 2 hours
  Decrease/increase in pressure for venous return measured by bedside continuous hemodynamic monitor supplied with continuous cardiac output monitoring with PiCCO(R) device
Change in resistance to venous return (dynes⋅sec⋅cm-5) | Baseline, every 5 minutes up to 30 minutes, 1 hour, 2 hours
  Decrease/increase in resistance te venous return measured by bedside continuous hemodynamic monitor supplied with continuous cardiac output monitoring with PiCCO(R) device
Change in systemic vascular resistance index (dynes⋅sec⋅cm-5) | Baseline, every 5 minutes up to 30 minutes, 1 hour, 2 hours
  Decrease/increase in systemic vascular resistance index measured by bedside continuous hemodynamic monitor supplied with continuous cardiac output monitoring with PiCCO(R) device
Change in venous return index (L/min/m2) | Baseline, every 5 minutes up to 30 minutes, 1 hour, 2 hours
  Decrease/increase in venous return index measured by bedside continuous hemodynamic monitor supplied with continuous cardiac output monitoring with PiCCO(R) device
Change in heart rate (bpm) | Baseline, every 5 minutes up to 30 minutes, 1 hour, 2 hours
  Decrease/increase in heart rate measured by bedside continuous hemodynamic monitor supplied with continuous cardiac output monitoring with PiCCO(R) device
Change in extra vascular lung water index (mL/kg) | Baseline and after 24 hours
  Decrease/increase in extra vascular lung water index measured with continuous cardiac output monitoring PiCCO(R) device
Change in global end diastolic volume index (mL/m2) | Baseline and after 24 hours
  Decrease/increase in global end diastolic volume index measured with continuous cardiac output monitoring PiCCO(R) device
Change in intrathoracic blood volume index (mL/m2) | Baseline and after 24 hours
  Decrease/increase in intrathoracic blood volume index measured with continuous cardiac output monitoring PiCCO(R) device
Creatinin (renal function) mmol/L | Baseline and after 24 hours
  Increase/decrease in creatinin (standard blood withdrawal within standard ICU treatment)
Electrolyte balance (potassium, sodium levels) (mmol/L) | Baseline and after 24 hours
  Increase/decrease in electrolyte balance (potassium, sodium levels) (standard blood withdrawal within standard ICU treatment)
Diuresis per hour (mL/hour) | Baseline, 1 hour, 2 hours and after 24 hours
  Increase/decrease in diuresis (standardly measured within standard ICU treatment)
Body weight (kg) | Baseline and after 24 hours
  Increase/decrease in body weight (standardly measured within standard ICU treatment)
Fluid balance (mL) | Baseline and after 24 hours
  Increase/decrease in fluid balance (mL) (standardly measured within standard ICU treatment)
Change in cardiac performance (eH) (dimensionless) | Baseline, every 5 minutes up to 30 minutes, 1 hour, 2 hours
  Increase/decrease in cardiac performance (eH)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Bakker, MD, PhD, Study Chair — Erasmus Medical Center
Locations (1):
- Catharina Hospital, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Under negotiable conditions sharing of data can be discussed.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Years
Access Criteria: Negotiable